CLINICAL TRIAL: NCT03081728
Title: Incidence Of Hemidiaphragmatic Paralysis With Patient Controlled Infusion Of Low Volume Of Ropivacaine After Usg Guided Low Dose Interscalene Brachial Plexus Block
Brief Title: Incidence Of Hemidiaphragmatic Paralysis After Usg Guided Low Dose Interscalene Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Pankaj, Junior resident, Department of Anaesthesia and Intensive Care, MD, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NK/3017/MD/051
Record Dates: First submitted 2017-03-12; First posted 2017-03-16 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Diclofenac; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Two groups: 1- block + GA 2- GA with multimodal analgesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- block (Experimental): will be given block and continuous infusion with bolus 10ml of 0.5% ropivacaine followed by infusion @ 2ml/hr of 0.2% ropivacaine
  Interventions: Device: Interscalene Block with Ropivacaine Hcl 0.2% Inj Vil 10Ml
- control (Experimental): IV analgesia only with diclofenac and paracetamol
  Interventions: Drug: IV diclofenac and IV paracetamol

INTERVENTIONS:
Device: Interscalene Block with Ropivacaine Hcl 0.2% Inj Vil 10Ml — bolus 10ml of 0.5% ropivacaine followed by infusion @ 2ml/hr of 0.2% ropivacaine
  Other Names: ROPIN
  Arms: block
Drug: IV diclofenac and IV paracetamol — iv diclofenac 75 mg TDS iv paracetamol 1gm TDS
  Other Names: vovran and perfalgan
  Arms: control

SUMMARY:
to put a catheter in interscalene brachial plexus USG guided and give a bolus of drug followed by 24 hours continous infusion of drug

DETAILED DESCRIPTION:
to put a catheter in interscalene brachial plexus USG guided and give a bolus of drug followed by 24 hours continous infusion of drug. To see hemidiaphragmatic paralysis by seeing diaphragmatic excursion on M mode Usg subcostal approach, to see post operative pain, patient satisfaction score, complications if any

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years and belonging to ASA grade I, II, III, undergoing either, shoulder surgery, (rotator cuff repair, acromioplasty, hemiarthroplasty, and total shoulder replacement) or surgery for proximal humerus fracture will be recruited for the study.

Exclusion Criteria:

* a) Patient refusal for interscalene block b) Severe respiratory disease (FEV1/FVC <0.7 and FEV1 < 80% of predicted) c) Allergy to amide local anaesthetic drugs d) Chronic opioid therapy e) Patients who cannot understand how to operate PCA and VAS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
incidence of hemidiaphragmatic paralysis | 24 hours
  incidence of hemidiaphragmatic paralysis by M mode USG to be seen

SECONDARY OUTCOMES:
postoperative pain | 24 hours
  VAS score will taken

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinha SK, Abrams JH, Barnett JT, Muller JG, Lahiri B, Bernstein BA, Weller RS. Decreasing the local anesthetic volume from 20 to 10 mL for ultrasound-guided interscalene block at the cricoid level does not reduce the incidence of hemidiaphragmatic paresis. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):17-20. doi: 10.1097/aap.0b013e3182030648. PMID 21751435
- [Background] Renes SH, Rettig HC, Gielen MJ, Wilder-Smith OH, van Geffen GJ. Ultrasound-guided low-dose interscalene brachial plexus block reduces the incidence of hemidiaphragmatic paresis. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):498-502. doi: 10.1097/AAP.0b013e3181b49256. PMID 19920426
- [Background] Fredrickson MJ, Price DJ. Analgesic effectiveness of ropivacaine 0.2% vs 0.4% via an ultrasound-guided C5-6 root/superior trunk perineural ambulatory catheter. Br J Anaesth. 2009 Sep;103(3):434-9. doi: 10.1093/bja/aep195. Epub 2009 Jul 16. PMID 19608563